CLINICAL TRIAL: NCT01469819
Title: The Effect of Lubiprostone on Transit Times Within the Alimentary Tract, Measured by Novel Smartpill Methodology in Patients With Chronic Constipation
Brief Title: Lubiprostone Effect on Gastrointestinal Tract Transit Times Measured by Smartpill in Patients With Chronic Constipation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Irene Sarosiek, Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUB-119
Record Dates: First submitted 2011-10-28; First posted 2011-11-10 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Chronic Idiopathic Constipation
Keywords: chronic constipation; constipation; idiopathic constipation; SmartPill; Wireless Motility Capsule; lubiprostone (Amitiza); small intestinal bacterial overgrowth
MeSH Terms: conditions — Constipation | interventions — Lubiprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lubiprostone (Experimental): Lubiprostone 24 mcg by mouth twice a day (BID) for 2 weeks.
  Interventions: Drug: Lubiprostone

INTERVENTIONS:
Drug: Lubiprostone — 24 mcg twice a day (BID) for 2 weeks.
  Other Names: Amitiza

SUMMARY:
The purpose of this study is to determine if lubiprostone may change the rate of movement of food and activities in the stomach and intestines in subjects whose gastrointestinal (GI) tract is slower due to constipation.

To be able to measure the time difference in the duration of transit of the FDA approved SmartPill capsule in all segments of gastrointestinal (GI) tract before and after exposure to lubiprostone.

The investigators anticipate to capture the possibility to reduce/eliminate the small intestinal bacterial overgrowth in chronically constipated patients after administration of study drug- lubiprostone.

DETAILED DESCRIPTION:
Lubiprostone is an effective treatment for chronic constipation. The mechanism of action of lubiprostone is through increasing fluid and mucus secretion and improving lubrication of the intestinal lumen. The effects of lubiprostone on gastrointestinal (GI) transit and small bacterial overgrowth (SIBO) have not been sufficiently explored.

The current study was designed to investigate whether: (a) lubiprostone alters GI transit and (b) affects SIBO in constipated patients.

Twenty nine female patients (mean age of 39 year: range 19-64) with chronic constipation received 2 weeks of lubiprostone (24 mcg b.i.d., P.O.). Stool consistency based on Bristol stool scale and the frequency of bowel movements were recorded. Gastric emptying time (GET), small bowel transit time (SBTT), colon transit time (CTT), combined small & large bowel transit time (SLBTT) and whole gut transit time (WGT) were measured using wireless motility capsule. Small bacterial overgrowth (SIBO) status was assessed by the lactulose breath test.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* At least a 6 months history of constipation. Constipation defined as follows:

  * Less than three complete spontaneous bowel movements per week and one or more of the following:

    1. At least 25% of stools are very hard and/or hard stools
    2. Sensation of incomplete evacuation following at least 25% of bowel movements.
    3. Straining on at least 25% of defecations. The above criteria are only applicable to spontaneous bowel movements. Patients who have no spontaneous bowel movements (bowel movements are preceded by laxative intake) are considered constipated and are eligible for this study.
* For patients ≥ 50 years of age, normal colonic anatomy as documented by colonoscopy, double-contrast barium enema, or flexible sigmoidoscopy performed within the previous 5 years.

Exclusion Criteria:

* Pregnancy or lactation.
* Subjects unwilling to practice adequate contraception throughout the period of screening through 14 days after the study termination.
* Use of laxatives 3 days immediately prior to randomization (except fiber or bulking agents).
* Use of any of the following drugs within 3 days prior to randomization:

  * Prokinetic agents (tegaserod, domperidone, cisapride, metoclopramide, erythromycin).
  * Medication containing opiates.
  * Anti-spasmodic (e.g., atropine, hyoscyamine, scopolamine, glycopyrrolate).
* Use of illegal drugs
* Regular consumption of 2 drinks of alcohol per day.
* Chronic nonsteroidal antiinflammatory drugs (NSAIDs) use
* Chronic use of H2 receptor antagonist or proton pump inhibitors (PPIs) within 14 days prior to screening.
* History of gastric or duodenal ulcer, inflammatory bowel disease(IBD), or chronic non-ulcer dyspepsia.
* Diabetes Mellitus (DM) type 1, Parkinson's disease.
* Existence of any medical condition that requires chronic therapy.
* Positive H. pylori serology
* Chronic active diverticulosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Sarosiek, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarosiek I, Bashashati M, Alvarez A, Hall M, Shankar N, Gomez Y, McCallum RW, Sarosiek J. Lubiprostone Accelerates Intestinal Transit and Alleviates Small Intestinal Bacterial Overgrowth in Patients With Chronic Constipation. Am J Med Sci. 2016 Sep;352(3):231-8. doi: 10.1016/j.amjms.2016.05.012. Epub 2016 May 24. PMID 27650225

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from University of Kansas Medical Center, in Kansas City, KS from July 2008 to August 2009. Additional participants were recruited from Texas Tech University Health Sciences Center - El Paso, in El Paso, TX between April 2012 and November 2012.
Pre-assignment Details: 37 participants recruited; 37 screened, 8 excluded. 25 of those subjects participated in small intestinal bacterial overgrowth (SIBO) testing and analysis.
Groups:
- All Participants: Due to the nature of this project, which did not include placebo, blinded portion of the investigation, all patients were exposed to study drug in a similar design. Lubiprostone 24 micrograms twice a day for 14 consecutive days was provided for qualified patients after all inclusionary criteria were met.
Period: Overall Study
Arm/Group | All Participants
Started | 37
Completed | 29
Not Completed | 8
Not completed — Withdrawal by Subject | 1
Not completed — Did not meet inclusionary criteria | 2
Not completed — Could not swallow SmartPill | 2
Not completed — Technical malfunction of SmartPill data | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 39 [19 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Time Reduction (Hours and Minutes) of Gastric Emptying (GE), Small Bowel (SB), Large Bowel (LB) and Whole Gut (WG) Transits Measured by SmartPill in Chronically Constipated Patients Before and After 2 Weeks of Therapy With Lubiprostone 24mcg Twice a Day.
Description: The change in transit time (TT), in hours and minutes, of gastric emptying (GE), small bowel (SB), large bowel (LB) and whole gut (WG) measured by SmartPill in 29 patients with chronic constipation after taking lubiprostone 24 micrograms twice a day (BID) for 2 weeks.
Time Frame: Measured at baseline and 2 weeks after baseline.
Measure: Mean (Standard Error); unit: Hours
Arm/Group | All Participants
Number analyzed (Participants) | 29
Hours
  Gastric Emptying Time before treatment | 7.0 (1.1)
  Small Bowel Transit Time before treatment | 5.9 (1.1)
  Small & Large Bowel Transit Time before treatment | 56.7 (8.7)
  Whole Gut Transit Time before treatment | 64.2 (8.5)
  Gastric Emptying Time after treatment | 9.3 (1.9)
  Small Bowel Transit Time after treatment | 4.5 (0.4)
  Small & Large Bowel Transit Time after treatment | 43.2 (4.6)
  Whole Gut Transit Time after treatment | 52.5 (4.8)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Changes in Number of Bowel Movements in Chronically Constipated Patients After 2 Weeks of Therapy With Lubiprostone 24mcg Twice a Day (BID).
Time Frame: Measured at baseline and 2 weeks after baseline
Measure: Mean (Standard Error); unit: number per week
Groups:
- All Participants: Due to the nature of this project, which did not include placebo, blinded portion to the investigation, all patients were exposed to study drug in a similar design. Lubiprostone 24 micrograms twice a day for 14 consecutive days was provided for qualified patients aster all inclusionary criteria were met.
Arm/Group | All Participants
Number analyzed (Participants) | 29
number per week
  Bowel Movements before treatment | 1.9 (0.1)
  Bowel Movements after treatment | 4.6 (0.4)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Changes in Time of GE, SB, LB and WG Transits Measured by SmartPill After 2 Weeks of Lubiprostone 24mcg BID in Chronically Constipated Patients.
Description: Changes in Time of GE, SB, LB and WG transits measured by SmartPill after 2 weeks of lubiprostone 24mcg BID in chronically constipated patients who increased stool frequency to ≥ 2 times increase per week vs. patients who increased stool frequency < 2 times increase per week.
Time Frame: Measured at baseline and 2 weeks after baseline.
Measure: Mean (Standard Error); unit: Hours
Groups:
- Responders: Subgroup of patients who clinically responded to lubiprostone defined as ≥ 2 times increase in their weekly bowel movement.
- Non-Responders: Subgroup of patients who had <2 times increase in their weekly bowel movement.
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 16 | 13
Hours
  Gastric Emptying Time before treatment | 9.6 (1.5) | 3.9 (1.2)
  Small Bowel Transit Time before treatment | 7.2 (2.1) | 4.5 (0.3)
  Small & Large Bowel Transit Time before treatment | 45.9 (6.8) | 70.1 (17.3)
  Whole Gut Transit Time before treatment | 55.5 (6.3) | 75.0 (17.3)
  Gastric Emptying Time after treatment | 11.6 (2.9) | 6.4 (2.1)
  Small Bowel Transit Time after treatment | 4.4 (0.6) | 4.5 (0.5)
  Small & Large Bowel Transit Time after treatment | 32.0 (4.3) | 57.0 (7.2)
  Whole Gut Transit Time after treatment | 43.7 (4.6) | 63.4 (8.5)
Statistical Analysis 1: Comparison: Responders vs Non-Responders; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Changes in Number of Bowel Movements Per Week Changes GE, SB, LB and WG Transit Times Measured by SmartPill in Chronically Constipated Patients Treated for 2 Weeks With Lubiprostone 24mcg Twice a Day.
Time Frame: Measured at baseline and 2 weeks after baseline.
Population: Number of Bowel Movements per week
Measure: Mean (Standard Error); unit: number per week
Groups:
- Responders: Subgroup of patients who clinically responded to lubiprostone defined as > 2 times increase in their weekly bowel movement compared to baseline.
Arm/Group | Responders | Non-Responders
Number analyzed (Participants) | 16 | 13
number per week
  Bowel Movements before treatment | 1.8 (0.1) | 2.1 (0.2)
  Bowel Movements after treatment | 6.0 (0.5) | 3.0 (0.2)
Statistical Analysis 1: Comparison: Responders vs Non-Responders; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Elimination of Small Intestine Bacterial Overgrowth (SIBO) in Chronically Constipated Patients Treated With Lubiprostone 24mcg Twice a Day for 2 Weeks.
Time Frame: Measured at baseline and 2 weeks after baseline.
Measure: Number; unit: participants
Groups:
- SIBO (+): Twenty-five patients were tested for SIBO before treatment with lubiprostone and 17 (68.0%) were SIBO (+) at baseline.
Arm/Group | SIBO (+)
Number analyzed (Participants) | 17
participants
  SIBO (+) participants before treatment | 17
  SIBO (+) participants after treatment | 10
  SIBO (+)→SIBO (-) participants after treatments | 7

ADVERSE EVENTS:
Groups:
- All Participants: Due to the nature of this project, which did not include placebo, blinded portion to the investigation, all patients were exposed to study drug in a similar design. Lubiprostone 24 micrograms twice a day for 14 consecutive days was provided for qualified patients after all inclusionary criteria were met.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 6/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=29)
Nausea (Gastrointestinal disorders) | 6 (6) — 6 patients experienced nausea after the drug administration of lubiprostone. Only 3 of these patients were diagnosed with prolonged gastric emptying time. None of these patients required any clinical attention or discontinuation of the study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No